CLINICAL TRIAL: NCT02032316
Title: URIPRENE: Feasibility Study to Evaluate the Preliminary Safety and Effectiveness of the Uriprene Stent Following Uncomplicated Ureteroscopy
Brief Title: Feasibility Study of the Uriprene Stent Following Uncomplicated Ureteroscopy
Acronym: URIPRENE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adva-Tec (Industry)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN 14-32-002
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Unilateral Ureteral Stone; Renal Stone Fragments ≤ 2mm
Keywords: Renal Stone; Ureteroscopy; Ureteral Stent; post-uncomplicated ureteroscopy; UURS
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional (Experimental): Placement of ureteral stent following post-ureteroscopy
  Interventions: Device: Post-Ureteroscopy ADVA-Tec Uriprene™ Degradable Temporary Ureteral Stent

INTERVENTIONS:
Device: Post-Ureteroscopy ADVA-Tec Uriprene™ Degradable Temporary Ureteral Stent — Renal stent placed after uncomplicated uteroscopy
  Other Names: Renal ureteral stent

SUMMARY:
A prospective, single-center, single-arm, trial to demonstrate safety and device performance of the ADVA-Tec Uriprene™ Degradable Temporary Ureteral Stent. This is a first-in-man clinical study in a small human population.

DETAILED DESCRIPTION:
Primary Objective: To assess the safety and feasibility of the Uriprene® Stent by assessing the time to complete degradation or the passage of stent fragments from the bladder by radiological assessment.

Subject Population: Patients with clinical symptoms consistent with unilateral ureteral or renal stone fragments ≤ 2mm, post-uncomplicated ureteroscopy (UURS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are > 18, < 80 years of age; inclusive of males and females.
2. Patients with unilateral ureteral or renal stone fragments < 2mm, post-uncomplicated ureteroscopy (UURS).
3. Patients with a height and body size able to accommodate a 20, 22, 24, 26, 28, or 30 mm long ureteral stent, as judged by the Investigator.
4. Patients with the ability to understand the requirements of the study, who have provided written informed consent, and who have agreed to return for the required follow-up assessments.

Exclusion Criteria:

1. Patients with a known contraindication for treatment with the Uriprene® Stent.
2. Patients with a history of an anatomical abnormality of the urinary tract.
3. Patients with a known upper or lower urinary tract infection at the time of stent insertion.
4. Patients with known renal insufficiency or chronic impairment.
5. Any condition, in the opinion of the investigator, in whom patients would not be eligible for treatment with the Uriprene® Stent.
6. Pregnant or lactating women, or women of childbearing potential who do not employ a reliable method of contraception as judged by the Investigator.
7. Patients who consume more than 14 drinks of alcohol per week (as this may affect degradation of the stent).
8. Presence of ureteral blockage or stricture
9. After failed guide wire placement or failed ureteroscopic access
10. Impacted ureteral stones still in place
11. Patients predisposed to urinary stasis e.g. neurogenic bladder, bladder outlet obstruction, known pregnancy
12. Patients with a solitary kidney
13. Presence of ureteral fistula
14. Presence of ureteral tumor
15. Presence of extrinsic compression of the ureter
16. Urinary tract infection
17. Staghorn calculi

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Safety | 90 days
  Composite of new-onset serious adverse event(s) including death, infection, the occurrence of surgery, re-hospitalization and or repeat hospitalization related to the device, or device related injury of the ureter.

SECONDARY OUTCOMES:
Technical Success | 90 days
  Technical success of the device defined as complete degradation of the stent within 90 days, as measured by radiology
Pain | 90 days
  Degree of comfort and pain as measured by the Pain, Symptom, and Satisfaction Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chew, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada